CLINICAL TRIAL: NCT05590923
Title: The Efficacy of Steroid-Sparing Anti-Emetic Therapy in Patients Treated With High or Moderate Emetogenic Chemotherapy; Single Center Non-Inferiority Open Label Randomized Controlled Trial
Brief Title: Steroid-sparing Therapy (Olanzapine) Versus Dexamethasone-based Therapy for Chemotherapy-induced Nausea and Vomiting
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped due to lower than expected accrual.
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2209-47
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to either the DEX group to receive dexamethasone or to the OLA group to receive olanzapine for the first cycle of chemotherapy.
  DEX group: dexamethasone (Decadron) 8 mg oral daily on days 2-4 after HEC (days 2-3 after MEC).
  OLA group: olanzapine (Zyprexa)10 mg oral each night on days 1-4 after HEC (days 2-3 after MEC).
  For the second cycle of chemotherapy, the subject will switch to the other group.
  Groups:
  OLA then DEX; DEX then OLA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OLA then crossover to DEX (Experimental): OLA group: olanzapine (Zyprexa) 10 mg oral each night after chemotherapy cycle 1 on days 1-4 after HEC (or days 1-3 after MEC).
  DEX group: dexamethasone (Decadron) 8 mg oral daily after chemotherapy cycle 2 on days 2-4 after HEC (or days 2-3 after MEC)
  Interventions: Drug: OLA group: Olanzapine; Drug: DEX group: Dexamethasone
- DEX then crossover to OLA (Active Comparator): DEX group: dexamethasone (Decadron) 8 mg oral daily after chemotherapy cycle 1 on days 2-4 after HEC (or days 2-3 after MEC)
  OLA group: olanzapine (Zyprexa) 10 mg oral each night after chemotherapy cycle 2 on days 1-4 after HEC (or days 1-3 after MEC).
  Interventions: Drug: OLA group: Olanzapine; Drug: DEX group: Dexamethasone

INTERVENTIONS:
Drug: OLA group: Olanzapine — OLA group: olanzapine 10 mg oral each night on days 1-4 after HEC (or days 1-3 after MEC).
  DEX group: dexamethasone (Decadron) 8 mg oral daily on days 2-4 after HEC (or days 2-3 after MEC).
  Other Names: Steroid-sparing therapy
Drug: DEX group: Dexamethasone — DEX group: dexamethasone (Decadron) 8 mg oral daily on days 2-4 after HEC (or days 2-3 after MEC)..
  OLA group: olanzapine 10 mg oral each night on days 1-4 after HEC (or days 1-3 after MEC).
  Other Names: Steroid therapy

SUMMARY:
The purpose of this research is to compare two drugs that are routinely used as standard of care for treating nausea and vomiting caused by chemotherapy. This study aims to see if the drug olanzapine is as good as the steroid drug dexamethasone for preventing nausea and vomiting after chemotherapy. Both drugs are listed as appropriate treatment options in the most recent version of National Comprehensive Cancer Network guidelines on Antiemesis.

DETAILED DESCRIPTION:
The study will include patients treated with high emetogenic chemotherapy (HEC) or moderate emetogenic chemotherapy (MEC). Emetogenic means that it may cause nausea and vomiting. Your participation will last for 2 cycles of chemotherapy.

For patients given high emetogenic chemotherapy (HEC):

As standard of care for nausea and vomiting after high emetogenic chemotherapy (HEC), subjects will receive fosaprepitant 150 mg IV once, palonosetron 0.25 mg IV once, dexamethasone 12 mg oral or IV once on day 1.

Patients will be randomly assigned to either the DEX group to receive dexamethasone or to the OLA group to receive olanzapine for the first cycle of chemotherapy.

1. DEX group: dexamethasone (Decadron) 8 mg oral daily on days 2-4.
2. OLA group: olanzapine (Zyprexa)10 mg oral each night on days 1-4. For the second cycle of chemotherapy, the subject will switch to the other group. For future cycles of chemotherapy, the subject will choose the drug that worked best.

For patients give moderate emetogenic chemotherapy (MEC):

As standard of care for nausea and vomiting after moderate emetogenic chemotherapy (MEC), subjects will receive granisetron 2 mg oral once and, dexamethasone 12 mg oral once on day 1.

Subjects will be randomly assigned to either the DEX group to receive dexamethasone or to the OLA group to receive olanzapine for the first cycle of chemotherapy.

1. DEX group: dexamethasone (Decadron) 8 mg oral daily on days 2-3.
2. OLA group: olanzapine (Zyprexa)10 mg oral each night on days 1-3. For the second cycle of chemotherapy, the subject will switch to the other group. For future cycles of chemotherapy, the subject will choose the drug that worked best.

Subjects (both HEC and MEC) will be asked to complete a survey prior to treatment on Day 1 of cycle 1 and cycle 2 prior to treatment. On Day 2 and Day 6 a member of the study will contact subjects by phone to complete another survey on any symptoms you may be experiencing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* confirmed cancer diagnosis
* starting cycle 1 of an FDA approved treatment that is categorized as high-emetogenic (nausea and vomiting inducing) chemotherapy per National Comprehensive Cancer Network® guidelines
* Eastern Cooperative Oncology Group performance score of 0 or 1
* appropriate renal function
* appropriate hepatic function
* appropriate hematologic function.

Exclusion Criteria:

* Patients will be excluded if they experience nausea or vomiting up to 24 hours before chemotherapy,
* currently on a glucocorticoid therapy
* contraindication to glucocorticoid therapy
* taking any medication that has antiemetic properties.
* scheduled or planned to receive radiation within one week of or concurrently with chemotherapy
* brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) over 120 hours following chemotherapy | 120 hours following chemotherapy
  Complete response (CR) over 120 hours following chemotherapy, where CR is the absence of emesis and no use of a rescue antiemetic medication, in the acute phase (<24 hours following chemotherapy), delayed phase (≥24 hours but ≤120 hours following chemotherapy) and overall (≤ 120 hours following chemotherapy).

SECONDARY OUTCOMES:
Complete control (CC- no emesis, no rescue medication and no more than minimal nausea) | 120 hours following chemotherapy
  no emesis, no rescue medication and no more than minimal nausea
Total Control (TC- no emesis, no rescue medication, no nausea) | 120 hours following chemotherapy
  no emesis, no rescue medication, no nausea
Severity of nausea and vomiting self-reported by patient questionnaire | 120 hours after chemotherapy
  None, mild or greater than mild
medication side effects | 120 hours after chemotherapy
  medication side effects including sedation, insomnia, agitation, indigestion/heartburn, depression, anorexia, increased appetite/hunger and rash/acne

CONTACTS AND LOCATIONS:
Overall Officials: Zane Waite, PharmD, BCOP, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No